CLINICAL TRIAL: NCT02964130
Title: A Multicenter Prospective Study on Failed Back Surgery Syndrome Pathway Optimization: A Focus on Patient Identification, Chronicization Factors and Outcome Predictors
Brief Title: Study on Failed Back Surgery Syndrome Pathway Optimization: A Focus on Patient Identification, Chronicization Factors and Outcome Predictors
Acronym: PREDIBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01144-47
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Failed Back Surgery Syndrome; Chronic Pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follow-up patient (Other): Medical follow-up visit
  Interventions: Other: No name

INTERVENTIONS:
Other: No name

SUMMARY:
This pilot study is part of a global project that aims to better define and understand features of FBSS/POPS "post-operative persistent syndrome patients (shortened as "FBSS" in the following project). FBSS is the acronym for Failed Back Surgery Syndrome, which has been defined as a chronic condition resulting from spinal interventions. Despite anatomically successful spine surgery, a significant proportion of patients is experiencing chronic refractory back and leg pain. In a recent multicentre study conducted on more than 100 refractory FBSS patients, (ESTIMET Study), the mean delay between pain occurrence and FBSS diagnosis was 5 years. Therefore, FBSS pattern and potential responder stratification might guide us to eventually develop a decision tool for identifying FBSS patients. Easing and helping diagnosis of FBSS should improve referral yield to specialists and accelerate patient flow through the care pathway. Hence, FBSS patients, who usually present a long standing history of pain, would have access to "appropriate" therapies earlier. This could lead to better outcomes. The aim of this multicentre, prospective study is to collect specific data that are not collected in routine in order to better define and understand the potential FBSS population and to accelerate the diagnostic and optimize the choice of appropriate treatment.

A multidisciplinary approach through a pain management clinical network, as it has been structured in Poitiers, will ensure that an exhaustive characterization of FBSS patients and their care pathway will be collected. In addition, since the cooperation between orthopaedic and neuro spine surgeons is not a common relationship found all over Europe (as it is observed in Poitiers), this study also aims to better understand the development of interactions between physicians/professionals and the substantial advantage which would result from bridging this gap. The N3MT (NeuroMapping Tools) software developed in Poitiers to collect data and assess objectively pain surface and intensity changes, before/after any treatment, with quantitative measurements, will be used as the central key of this project.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated the Informed Consent Form.
* Patient is ≥ 18 years of age at time of "Informed Consent Form" signature.
* Patient had most recent back surgery more than 6 months ago.
* Patient has developed post-operative Chronic Back with or without Leg Pain (potential FBSS).
* Patient has persistent back pain for more than 6 months.
* Average low back or leg pain is ≥ 4 as assessed by the baseline NPRS.

Exclusion Criteria:

* Patient has already a confirmed FBSS diagnosis.
* Patient is or has been treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system.
* Investigator suspects substance abuse that might confound the study results.
* Patient has a life expectancy of less than 12 months beyond study enrollment.
* Patient is less than 18 years of age.
* Patient is pregnant or planning to become pregnant during the course of the study.
* Patient is unable to undergo study assessments or complete questionnaires independently (e.g., is illiterate).
* Patient is a member of a vulnerable population.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical diagnosis of FBSS | 12 month-follow up visit
  Incidence of clinical diagnosis of FBSS in the broad population of post-surgical pain syndrome, identified by multidisciplinary team of independent experts (1 pain physician, 1 neurosurgeon and 1 psychiatric), with morphological and clinical characterization of the syndrome.

SECONDARY OUTCOMES:
Pain intensity (NRPS) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
  * Reduction of the NRPS score measuring pain intensity: Global pain, Back pain and Leg pain.
  * Proportion of patients with NRPS score < 4.
  * Proportion of patients obtaining a reduction ≥ 25%, 50% and 75%: Global pain, Back pain and Leg pain NRPS.
Pain surface and intensity (Mapping Tool) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
  * Reduction of the Global Pain Surface measured on the NeuroPain't module of the software, during treatment, before/after a therapeutic strategy is used.
  * Reduction of pain intensities associated with the quantitative surface measurements.
  * Reduction of the mechanical/neuropathic component of objective pain.
Functional capacity (ODI) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
Quality of life (EQ5D) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
Psychological State (HADS) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
Pain Catastrophizing Scale (PCS CF) | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits
Adverse Events/ Serious Adverse Events | Initial visit and 3 month, 6 month, 9 month and 12 month-follow up Visits

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RIGOARD, PU-PH, Principal Investigator — Poitiers Hospital University
Locations (1):
- Poitiers Hospital University, Poitiers, France

REFERENCES:
- [Derived] Billot M, Ounajim A, Moens M, Goudman L, Deneuville JP, Roulaud M, Nivole K, Many M, Baron S, Lorgeoux B, Bouche B, Lampert L, David R, Rigoard P. The Added Value of Digital Body Chart Pain Surface Assessment as an Objective Biomarker: Multicohort Study. J Med Internet Res. 2025 Apr 16;27:e62786. doi: 10.2196/62786. PMID 40239206